CLINICAL TRIAL: NCT06191575
Title: A Pilot Study of 7 Tesla MRI Neuroimaging in Testicular Cancer Patients With Hypogonadism and Androgen Replacement Therapy
Brief Title: 7 Tesla MRI Neuroimaging in Testicular Cancer Patients With Hypogonadism and on Androgen Replacement Therapy
Status: Suspended | Type: Observational
Why Stopped: Study team is conducting interim analysis.
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4T-22-1; NCI-2022-07931 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4T-22-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hypogonadism; Malignant Testicular Germ Cell Tumor
MeSH Terms: conditions — Hypogonadism; Testicular Neoplasms | interventions — Specimen Handling; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (7T MRI, cognitive assessment, blood collection): Patients undergo 7T MRI over 1-2 hours at baseline and at 12 months after baseline. Patients also undergo a proctored cognitive assessment over approximately 1 hour prior to each MRI. Additionally, patients undergo blood sample collection at screening and at 12 months after baseline MRI.
  Interventions: Procedure: 7 Tesla Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Cognitive Assessment

INTERVENTIONS:
Procedure: 7 Tesla Magnetic Resonance Imaging — Undergo 7T MRI
  Other Names: 7 T MRI; 7 Tesla MRI
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cognitive Assessment — Undergo cognitive assessment

SUMMARY:
This study evaluates 7 Tesla (T) magnetic resonance imaging (MRI) in observing changes in the brain (neuroimaging) in testicular cancer patients who have decreased testosterone (hypogonadism) and are on testosterone (androgen) replacement therapy. Symptoms of hypogonadism can include fatigue, weakness, loss of libido, depression, poor concentration and erectile dysfunction. Some patients experience mental changes after diagnosis and treatment. There is some evidence that hypogonadism produces structural changes in the brain. The 7T MRI uses radio waves and a very powerful magnet linked to a computer to create detailed pictures of areas inside the body. This study may help researchers learn if 7T MRI can produce better images to assess the changes in the brain structure of testicular patients with hypogonadism and on androgen replacement therapy (ART).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess longitudinal structural changes in brain architecture using MRI in hypogonadal men with testis cancer being treated with androgen replacement therapy.

OUTLINE: This is an observational study.

Patients undergo 7T MRI over 1-2 hours at baseline and at 12 months after baseline. Patients also undergo a proctored cognitive assessment over approximately 1 hour prior to each MRI. Additionally, patients undergo blood sample collection at screening and at 12 months after baseline MRI.

ELIGIBILITY:
Inclusion Criteria:

* Males age >= 18 years
* Diagnosed with germ cell tumor of the testis (seminoma or non-seminoma) and treated with radical orchiectomy
* Diagnosed with hypogonadism and started androgen replacement therapy 6 months prior (+/- 2 weeks)
* Ability to understand and the willingness to sign a written informed consent
* Ability to undergo imaging procedure without any form of sedation

Exclusion Criteria:

* History of any neuropsychiatric disease
* History of narcotic use or psychiatric medications
* History of ART prior to current ART regimen
* Standard contraindications for MRI:

  * Prior work as a machinist or metal worker, or history of metal being removed from the eyes
  * Cardiac pacemaker or internal pacing wires
  * Non-MRI compatible vena cava filter, vascular aneurysm clip, heart valve, spinal or ventricular shunt, optic implant, neuro-stimulator unit, ocular implant, or intrauterine device, or
  * Claustrophobia, or uncontrollable motion disorder
* Current active second malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male testicular patients with hypogonadism on androgen replacement therapy recruited from University of Southern California/Kenneth Norris, Jr Comprehensive Cancer Center and Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain structural connectivity | At baseline and 12 months
  Measured using T1-weighted and diffusion tensor magnetic resonance imaging (MRI).
Brain functional connectivity | At baseline and 12 months
  Measured using resting-state functional MRI.
Brain metabolic profiles | At baseline and 12 months
  Evaluated by MR spectroscopy.
Brain perfusion | At baseline and 12 months
  Evaluated by arterial spin labeling MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Shiroishi, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California